CLINICAL TRIAL: NCT03500653
Title: Curcumin Supplementation as an Add on Treatment for Patients With Inflammatory Bowel Diseases Treated With Vedolizumab
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henit Yanai (Other)
Collaborators: Shaare Zedek Medical Center (Other)
Responsible Party: Sponsor-Investigator, Henit Yanai, Head of IBD center, Rabin Medical Center
Organization: Rabin Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RMC-0290-17
Record Dates: First submitted 2017-06-14; First posted 2018-04-18 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Curcumin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Active Comparator): 4 gr Curcumin daily for 1 year in addition to vedolizumab 300 mg per infusion (standard of care)
  Interventions: Dietary Supplement: Curcumin
- Sham (Placebo Comparator): 4 gr placebo daily for 1 year in addition to vedolizumab300 mg per infusion (standard of care)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Curcumin — 4 gr curcumin
  Arms: Active
Dietary Supplement: Placebo — 4 gr placebo
  Arms: Sham

SUMMARY:
Introduction: The pathogenesis of inflammatory bowel diseases (IBD) is characterized by dysregulation of the innate immune response it's associated with Th1, Th17 up-regulation, reflected by increased cytokine secretion including TNF-α. A main effective therapeutic interventions is blocking TNFα. Vedolizumab, an anti integrin, is a new class of treatment designed to block trafficking of lymphocytes in the gut. Clinical trials and real life experience response rates at week 6 range between 30-45%. Curcumin suppresses NFκβ levels via alteration of TLR2/4 pathways lowering TNF-α upstream. Curcumin is safe and efficacious in inducing response and remission in mild-moderate Ulcerative colitis (UC) and maintaining remission when used as an add-on to 5ASA derivatives, only with strict adherence to treatment overtime.

Objectives: Facing the low rate of response to therapies in IBD, the need for new treatments and the use of combination strategies lead us to believe that combining vedolizumab and curcumin may have a synergistic effect and will enable optimal immunomodulation.

Hypothesis: Concomitant oral curcumin in IBD patients with colonic involvement will augment remission rates as well as clinical and biochemical response.

Type of research and methods of data collection: A randomized controlled trial in 84 adults with colonic IBD (UC and CD). Eligible patients are during vedolizumab induction, patients will randomized will be into curcumin or placebo. Data will managed by investigators.

ELIGIBILITY:
Inclusion Criteria:

1. Established inflammatory bowel disease
2. Age ≥18 years old
3. At inclusion all patients must have a documented active colonic involvement based on either endoscopy or imaging:
4. Commencing vedolizumab therapy according to the treating physician or on active therapy up to 6-weeks.
5. Active luminal disease:

   CD- HBI ≥325, 26 UC- partial Mayo ≥227
6. Evident active disease on endoscopy or imaging within 2-week from inclusion or elevated inflammatory markers at screening (CRP> 0.5 mg/dl, or fecal calprotectin>100 μgr/gr stool or ESR >40).

Exclusion Criteria:

1. CD- isolated small bowel disease (L1) UC- proctitis (E1)
2. Perianal disease
3. Pregnancy
4. Biliary obstruction
5. Concomitant treatment with beta blockers, anti-coagulants, and norfloxacin (relative contra indications to curcumin therapy).
6. Curcumin supplementations within the last 6 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-06-09 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Clinical remission- Crohn's disease patients | 52 weeks
  Crohn's disease patients - disease activity indexe: Harvey Bradshow index (HBI) less that 3
Clinical remission- ulcerative colitis patients | 52 weeks
  Disease activity index - partial Mayo score less than 2

SECONDARY OUTCOMES:
Disease response- Crohn's disease patients | 52 weeks
  Disease activity index- Harvey Bradshow index (HBI ) a drop of 3 points
Disease response- ulcerative colitis patients | 52 weeks
  Disease activity index -partial Mayo score a drop of 2 points
Biochemical remission | 52 weeks
  Fecal calprotectin less than 150 µg/gr
Biochemical remission | 52 weeks
  C reactive protein (CRP) less thn 0.5 mg/dl

CONTACTS AND LOCATIONS:
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: Undecided